CLINICAL TRIAL: NCT06318325
Title: Growth Process and Development of Muscle, Bone, and Tendon in Correlation With Injuries in Young Gymnasts During Adolescence
Brief Title: Growth Process and Development of the Musculoskeletal System in Young Gymnasts
Status: Completed | Type: Observational
Sponsor: University of Haifa (Other)
Collaborators: The Academic college Levinsky-Wingate at the Wingate Institute, Netanya, Israel (Unknown)
Responsible Party: Principal Investigator, Gali Dar, PHD, Prof., University of Haifa
Other Study IDs: ADINEGEV-2021_102
Record Dates: First submitted 2024-03-12; First posted 2024-03-19 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Development, Adolescent
Keywords: musculoskeletal; menarche; athlete
MeSH Terms: interventions — Physical Examination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- gymnasts: gymnasts ages 9-16 years. All participants are of competitive level, each participating in at least four competitions per year
  Interventions: Diagnostic Test: examination

INTERVENTIONS:
Diagnostic Test: examination — examination of tendon, muscle joints and injuries

SUMMARY:
assessment of the musculoskeletal system will be performed twice a year, for three years of young gymnasts.

DETAILED DESCRIPTION:
Aims: To examine the changes in the anatomical and morphological features in the skeleton of young female artistic and rhythmic gymnasts and follow the risk of injuries during the period of pubertal growth.

Methods: 200 gymnasts (100 rhythmic and 100 artistic) will participate. Measurements will be performed at the beginning and the end of each year, for three years. Each gymnast will be examined for the following: asked about her menarche, assessed by a physician for Tanner stages, and will answer the Triad-specific self-report questionnaire. Anthropometric measurements (height, weight, BMI), muscle strength (using hand-held dynamometer), joint range of motion (using goniometer), scoliosis, and Beighton test for hypermobility will be assessed. In addition, the gymnasts will be scanned by using three different ultrasounds: Bone age for the skeletal age, SOS for the bone properties, and ultrasound tissue characterization for the tendon structure. The gymnasts will be asked about their physical training history, frequency, and training intensity. Each gymnast will be asked whether she had pain or injuries during the period she has been training, as well as a physical and injuries evaluation that will be conducted by a physician.

Once a month a telephone follow-up with the trainer regarding any pain or injuries in the last month will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* training at least 4 times per week,
* a minimum of 16 hours per week, at a competitive level.
* The gymnasts exercised fully three months before the beginning of the study
* have not been absent more than three days from training due to pain, discomfort, or injury.

Exclusion Criteria:

* present injury causing pain
* missing training.

Ages: 9 Years to 16 Years | Sex: Female
Age Groups: Child
Gender Based: Yes — young female gymnasts
Study Population: young female gymnasts training on a regular basis and competitive level
Sampling Method: Non-Probability Sample
Enrollment: 274 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-12-15 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
ultrasound tissue characterized | baseline, twice a year for 3 years
  percentage of type 1,2,3,4 fibers within the tendon
muscle strength test | baseline, twice a year for 3 years
  hand held dynamometer assessment of ankle, knee and hip muscles
range of motion | baseline, twice a year for 3 years
  goniometer assessment for lower extremities joints
bone strength | baseline, twice a year for 3 years
  tibia bone strength assessment using Sunlight MiniOmni Ultrasound Bone Sonometer
Bone Age | baseline, twice a year for 3 years
  bone age of the radius bone using ultrasound for bone age

CONTACTS AND LOCATIONS:
Overall Officials: Gali Dar, Principal Investigator — University of Haifa
Locations (1):
- The Academic college Levinsky-Wingate at the Wingate Institute, Netanya, Israel

IPD SHARING:
Plan to Share IPD: Undecided